CLINICAL TRIAL: NCT00320073
Title: A Two Arm Phase I Dose Escalation Trial of Vinflunine With Erlotinib or Pemetrexed in Refractory Solid Tumors
Brief Title: Vinflunine and Erlotinib or Pemetrexed in Treating Patients With Unresectable or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0509; CDR0000550148 (Other: PDQ number)
Record Dates: First submitted 2006-04-27; First posted 2006-05-03 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Erlotinib Hydrochloride; Pemetrexed; vinflunine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Pemetrexed, Vinflunine, Folate, B12, Dexamethasone, Ondansetron, Midazolam
  Interventions: Drug: pemetrexed disodium; Drug: vinflunine
- Arm B (Experimental): Vinflunine, Erlotinib, Ondansetron, Midazolam
  Interventions: Drug: erlotinib hydrochloride; Drug: vinflunine

INTERVENTIONS:
Drug: erlotinib hydrochloride — 75 mg to 150mg
  Arms: Arm B
Drug: pemetrexed disodium — Pemetrexed is administered intravenously over 10 minutes, every 21 days
  Arms: Arm A
Drug: vinflunine — Vinflunine is administered intravenously over 20 minutes and should be given after pemetrexed, every 21 days

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as vinflunine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Erlotinib and pemetrexed may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving vinflunine together with erlotinib or pemetrexed may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of vinflunine when given together with erlotinib or pemetrexed in treating patients with unresectable or metastatic solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Define the maximum tolerated dose (MTD) of vinflunine and pemetrexed disodium in patients with unresectable or metastatic solid tumors.
* Define the MTD of vinflunine and erlotinib hydrochloride in these patients.

Secondary

* Determine the preliminary safety and efficacy (reported descriptively per patient response; tumor specific response rate reported if applicable) of these regimens.
* Correlate CYP3A4 activity, as measured by midazolam clearance, with vinflunine plasma clearance.

OUTLINE: This is a nonrandomized, open-label, dose-escalation study. Patients are assigned to 1 of 2 treatment groups.

* Group 1: Patients receive pemetrexed disodium IV over 10 minutes and vinflunine IV over 20 minutes on day 1.

Cohorts of 3-6 patients receive escalating doses of pemetrexed disodium and vinflunine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Additional patients may be treated at the MTD.

* Group 2: Patients receive vinflunine IV over 20 minutes on day 1 and oral erlotinib hydrochloride once daily on days 2-21 of course 1 and on days 1-21 of all subsequent courses.

Cohorts of 3-6 patients receive escalating doses of erlotinib hydrochloride and vinflunine until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Additional patients may be treated at the MTD.

In both groups, courses repeat every 21 days in the absence of unacceptable toxicity.

Blood samples are collected on day 1 of course 1 for pharmacodynamic studies.

After completion of study treatment, patients are followed for 30-40 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumors

  * Advanced/unresectable or metastatic disease
* Refractory to standard therapy OR no standard therapy exists
* No lymphoma
* Measurable or evaluable disease

  * Measurable disease is defined as at least one target lesion measuring ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan
  * Evaluable disease includes ascites, pleural effusion, bone metastases, pulmonary lymphangitic spread, and lesions not meeting above criteria as measurable

    * Patients with clinically significant ascites or pleural effusions that cannot be controlled by drainage are not eligible
* Brain metastases allowed if CNS-directed treatment has been given, patient has been off CNS-directed therapy for > 3 months, and CNS disease has been clinically and radiographically stable for at least 8 weeks

PATIENT CHARACTERISTICS:

* Life expectancy > 3 months
* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Creatinine clearance ≥ 60 mL/min

  * Patients assigned to group 1 with creatinine clearance 45-80 mL/min must be able to withhold NSAIDS during pemetrexed disodium administration
* Total bilirubin ≤ 1.5 mg/dL
* AST and ALT ≤ 3 times upper limit of normal (ULN) OR ≤ 5 times ULN if due to known liver metastases
* No New York Heart Association class III or IV heart failure
* No unstable angina
* No myocardial infarction within the past 6 months
* No poorly controlled hypertension
* No prior allergic reaction to any vinca alkaloid
* No uncontrolled active infection or severe illness
* Able to receive vitamin B12 and folate supplementation and dexamethasone during chemotherapy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after last dose of chemotherapy

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior chemotherapy, investigational agents, or surgery
* Concurrent cytochrome P450/CYP3A4 inducers or inhibitors are allowed provided patient has been on a stable dose for ≥ 2 weeks prior to study entry
* No concurrent ketoconazole, itraconazole, ritonavir, amprenavir, or indinavir
* No concurrent enzyme-inducing antiepileptic drugs (EIAEDs) (e.g., phenytoin, carbamazepine, phenobarbital, primidone, or oxcarbazepine) for patients assigned to group 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-08; Primary Completion 2008-10 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of vinflunine and pemetrexed disodium | 1 year
  The MTD is defined as the dose cohort where approximately 0.20 of patients experience DLT. Standard "groups of three" phase I dose escalation design will be used in each arm. Each dose cohort will accrue a minimum of three patients.The estimated MTD is the dose level below the dose that induced dose limiting toxicity (DLT) in one third or more of patients
Maximum tolerated dose (MTD) of vinflunine and continuously dosed erlotinib | 1 year
  The MTD is defined as the dose cohort where approximately 0.20 of patients experience DLT. Standard "groups of three" phase I dose escalation design will be used in each arm. Each dose cohort will accrue a minimum of three patients.The estimated MTD is the dose level below the dose that induced dose limiting toxicity (DLT) in one third or more of patients
Maximum tolerated dose (MTD) of vinflunine and intermittently dosed erlotinib | 1 year
  The MTD is defined as the dose cohort where approximately 0.20 of patients experience DLT. Standard "groups of three" phase I dose escalation design will be used in each arm. Each dose cohort will accrue a minimum of three patients.The estimated MTD is the dose level below the dose that induced dose limiting toxicity (DLT) in one third or more of patients

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth C. Dees, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States